CLINICAL TRIAL: NCT07067463
Title: A Phase 3, Randomized, Double-blind, Efficacy and Safety Study Comparing Orelabrutinib to Placebo in Patients With Primary Progressive Multiple Sclerosis
Brief Title: A Study of Orelabrutinib in Patients With Primary Progressive Multiple Sclerosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zenas BioPharma (USA), LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZB020-03-001
Record Dates: First submitted 2025-07-03; First posted 2025-07-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis (MS) Primary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — orelabrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orelabrutinib Group (Experimental)
  Interventions: Drug: Orelabrutinib
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orelabrutinib — Orally
  Arms: Orelabrutinib Group
Drug: Placebo — Orally
  Arms: Placebo Group

SUMMARY:
Orelabrutinib is a CNS-penetrable BTK inhibitor. This is a phase 3, randomized, double-blind, parallel-group, multicenter study to evaluate the efficacy and safety of orelabrutinib compared with placebo in patients with PPMS. Patients will be treated for approximately 30 to 60 months, with a minimum treatment duration of 12 months. The study will enroll approximately 705 subjects in a 2:1 randomization (orelabrutinib: placebo), globally.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age, inclusive
* Diagnosed with Primary Progressive MS (PPMS) according to 2017 McDonald criteria
* Participant must have documented evidence of disability progression observed during the 24 months before screening.
* Expanded disability status scale (EDSS) score between 3.0 to 6.5 points, inclusive, at Screening.

Exclusion Criteria:

* Diagnosed with relapsing-remitting MS (RRMS) or secondary progressive MS (SPMS)
* Immunologic disorder other than MS or any other conditions requiring oral, intravenous (IV), intramuscular, or intra-articular corticosteroid therapy.
* History or current diagnosis of other neurological disorders that may mimic MS
* History of any other significant active medical condition
* History of suicidal behavior within 6 months prior to Screening
* Any prior history of malignancy if no recurrence within 5 years
* Patients on anticoagulation, or antiplatelet therapy will be excluded
* Patients took strong/moderate CYP3A inhibitors or strong/moderate CYP3A inducerswithin 14 days
* Clinically significant laboratory abnormalities at Screening.
* Any allergy, contraindication, or inability to tolerate orelabrutinib or any of the excipients in the study intervention
* Vaccination with live or live-attenuated virus vaccine within 1 month prior to Screening
* History of alcohol abuse or alcohol use disorder or other drug abuse within 12 months prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 705 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Time to onset of composite confirmed disability progression (cCDP) , confirmed over at least 12 weeks (12-week cCDP) | Up to approximately 120 weeks
  * Expanded disability status scale (EDSS) score increase ≥ 1.0 point from baseline when the baseline score is ≤ 5.0, or ≥ 0.5 points from baseline when the baseline score is > 5.0, OR
  * ≥ 20% increase in the Timed 25-Foot Walk Test (T25FWT), OR
  * ≥ 20% increase in the 9-hole Peg Test (9HPT)

SECONDARY OUTCOMES:
Time to onset of composite confirmed disability progression (cCDP) , confirmed over at least 24 weeks (24-week cCDP) | Up to approximately 120 weeks
Time to onset of confirmed disability progression (CDP) , confirmed over at least 24 weeks (24-week CDP) | Up to approximately 120 weeks
  Expanded disability status scale (EDSS) score increase ≥ 1.0 point from baseline when the baseline score is ≤ 5.0, or ≥ 0.5 points from baseline when the baseline score is > 5.0.
MRI T2 lesion | Up to approximately 120 weeks
  The total number of new/enlarging T2 lesions on MRI scans of the brain from baseline to Week 120
12-week CDP | Up to approximately 120 weeks
  Time to onset of CDP, confirmed over at least 12 weeks
Time to onset of CDP defined as ≥ 20% increase on 9-hole Peg Test (9HPT) from baseline, confirmed over at least 12 weeks (12-week CDP-9HPT) | Up to approximately 120 weeks
Time to onset of CDP defined as ≥ 20% increase on Timed 25-Foot Walk Test (T25FWT) from baseline, confirmed over at least 12 weeks (12-week CDP-T25FWT) | Up to approximately 120 weeks
24-week cCDI | Up to approximately 120 weeks
  Time to onset of composite confirmed disability improvement (cCDI) events, confirmed over at least 24 weeks
24-week CDI-9HPT | Up to approximately 120 weeks
  Time to onset of CDI on 9HPT defined as ≥ 20% decrease on the 9HPT score from baseline, confirmed over at least 24 weeks
24-week CDI | Up to approximately 120 weeks
  Time to onset of CDI on EDSS confirmed over at least 24 weeks
24-week CDI-T25FWT | Up to approximately 120 weeks
  Time to onset of CDI on T25FWT defined as ≥ 20% decrease on the T25FWT score from baseline, confirmed over at least 24 weeks
SDMT | Up to approximately 120 weeks
  The change in cognitive function as assessed by Symbol Digit Modalities Test (SDMT)
AEs | Up to approximately 120 weeks
  Safety as assessed by the nature, severity, and incidence of adverse events (AEs) (graded according to National Cancer Institute-Common Terminology Criteria for AEs, NCI-CTCAE version 5.0); vital signs; electrocardiograms (ECGs); and clinical laboratory safety parameter

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Neurology Associates, PA, Maitland, Florida
  - Premier Neurology, Greenville, South Carolina